CLINICAL TRIAL: NCT02424266
Title: Three Dimension Tomography of Eye Structures by White Light Imaging Device
Acronym: 3D-WLT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Avner Belkin, MD, Meir Medical Center
Other Study IDs: MMC-0166-13
Record Dates: First submitted 2015-04-01; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Healthy Subjects; Moderate to Severe Keratoconjunctivitis Sicca (KCS); Dry Eye Syndrome (DES)
Keywords: Tear film; Imaging; Tomogrophy; dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy subjects: None invasive imaging of the tear film for subjects with no eye disease
  Interventions: Device: None invasive imaging of the tear film (AdOM)
- keratoconjunctivits sicca (KCS) and Dry Eye Syndrome (DES): None invasive imaging of the tear film for KCS and DES patients as confirmed by a cornea specialist
  Interventions: Device: None invasive imaging of the tear film (AdOM)

INTERVENTIONS:
Device: None invasive imaging of the tear film (AdOM) — White light tomography imaging

SUMMARY:
The purpose of this study is to investigate the ability of an imaging device, developed by AdOM Advanced Optical Technologies Ltd. ("AdOM"). The device allows a three-dimensional imaging of the ocular tissues, specifically the tear film layers and the retinal layers. The device is based on the use of white light.

In this initial study, the device will be used to assess the tear film which coats the corneal surface in healthy subjects as well as in moderate-to-severe Keratoconjunctivitis Sicca (KCS) or Dry Eye Syndrome (DES). The ability of the device to assess the retinal layers will be evaluated in the second phase of the study.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the ability of an imaging device, developed by AdOM Advanced Optical Technologies Ltd. ("AdOM"). AdOM has produced an imaging device based on a standard fundus camera that uses white light, and as combined with new algorithms allows for a new reconstruction of three-dimensional images. The materials from which the Medical Instrumentation and Device are comprised are optical components (lenses), a broadband light source power, mechanical engines, beam splitters, and optical filters. The device will in addition contain camera sensors and a spectral detector. These elements are linked to a computer which includes control software and a user interface. The device allows a three-dimensional imaging of the ocular tissues, specifically the tear film layers and the retinal layers.

In this initial study, the device will be used to assess the tear film which coats the corneal surface in healthy subjects as well as in moderate-to-severe Keratoconjunctivitis Sicca (KCS) or Dry Eye Syndrome (DES). The ability of the device to assess the retinal layers will be evaluated in the second phase of the study.

The aqueous layer of the tear layer thickness is expected to be measured at an accuracy level of approximately one nanometer. All values will be measured over time and thus it will be possible to deduce the breakup time of the tear layer and the evaporation rate. It is possible that information will also be provided on the mucin layer and its level of sharpness.

Using the device will include the following steps:

1. Resting the head and fixing it with the assistance of the chin and forehead rests.
2. Locating and focusing the device on the cornea or retina with the help of the examiner.
3. Identifying the retinal and vitreous layers and pressing to start measurement or, alternatively:
4. Identifying the tear film layers and pressing to start the measurement.
5. Pressing on the button to end the measurement. The expected measurement duration is 20 to 70 seconds. Analysis of the returned light will describe at each second the thickness of the layers and the continuity of the surface.

Study population:

A total of 20 healthy patients. A total of 40 adult male or female patients with moderate-to-severe KCS or DES.

Conduct of the Study:

This is a case-control, non-randomized observational study. The study will include two visits: a screening visit and a study visit.

During the screening visit the patients will sign the informed consent form and a full medical history will be recorded. All ocular signs and symptoms will be evaluated and a full biomicroscopic examination will be performed. Disease activity will be assessed using the Dry Eye Symptom Score (DESS), Schirmer Test (ST), tear meniscus height (TM), tear break-up time (BUT), and fluorescein staining (FS).

The second visit will be scheduled up to 4 weeks after the screening visit. During the second visit (the photography session), all ocular signs and symptoms will be evaluated and a full biomicroscopic examination will be performed. Disease activity will be assessed using the Dry Eye Symptom Score (DESS), Schirmer Test (ST), tear meniscus height (TM), tear break-up time (BUT), and fluorescein staining (FS).

The tear film layer will be photographed by the investigational device and the participation of the volunteers in the study will end with the end of the photography session.

Time frame: participants will be followed for the duration of their participation in the study which is expected to be up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

Age >/= 18 years Healthy controls - without dry eyes

Patients with a diagnosis of moderate-to-severe KCS as defined by all of the following:

1. The presence of at least one ocular symptom of dryness scored at > 2 (where 0 = none and 4 = very severe /interferes with normal activities)
2. Positive Schirmer test (ST without anesthesia) < 7 mm/5 min in either eye
3. Positive fluorescein stainig (FS), defined as a corneal punctate fluorescein staining score of > 1 in either eye, where 0 = none and 3 = severe.

Exclusion Criteria:

1. Stevens-Johnson Syndrome
2. Post-burn ocular injury
3. Chronic ocular disease other than KCS requiring topical treatment
4. Ocular herpes simplex virus infection
5. Use of contact lenses
6. Persistent Intraocular Inflammation or Infection
7. Active blepharitis of greater than mild degree
8. Recent surgical occlusion of the lacrimal puncta
9. Subepithelial cornea scarring
10. Anesthetic or neurotrophic corneas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 healthy subject with no ocular disease 40 subjects with moderate to severe keratoconjunctivitis sicca or dry eye syndrome
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Safety (Ocular symptoms) | One month
  Ocular symptoms, including - I. pain (graded as 0-none, 1- mild discomfort, 2-moderate pain, 3- severe pain, 4- very severe), II. burning (graded as 0-none, 1- mild , 2-moderate, 3- severe, 4- very severe), itching (graded as 0-none, 1- mild , 2-moderate, 3- severe, 4-very severe) 2. Red eye (graded as 0-none, 1- mild , 2-moderate, 3- severe, 4- very severe)

SECONDARY OUTCOMES:
Imaging capabilities (field of view, resolution) | On sight
  1. field of view, measured in millimeters
  2. resolution measured in line per millimeters
Tear film measurements (lipid layer thickness, aqueous layer thickness) | on sight
  1. lipid layer thickness measured in microns
  2. aqueous layer thickness measured in microns

CONTACTS AND LOCATIONS:
Overall Officials: Noa Geffen, MD, Principal Investigator — Meir Medical Center